CLINICAL TRIAL: NCT01604798
Title: Serum Proteomic Profiling for the Early Diagnosis of Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Professor of General Surgery, Fudan University
Other Study IDs: ZSCG-001; 30973416 (Other Grant/Funding Number: the National Natural Science Foundation)
Record Dates: First submitted 2012-05-17; First posted 2012-05-24 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Colorectal Neoplasms
Keywords: proteomics; serum peptides; colorectal cancer; MALDI-TOF MS
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All fasting blood samples were prepared without anticoagulant and left to clot at room temperature for 1.5 h. The serum was then isolated by centrifugation at 3000 g for 10 min at room temperature and stored at -80℃. All samples were subjected to one freeze-thaw cycle.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Colorectal Cancer Patients: Patients with histologically confirmed colorectal cancer
  Interventions: Other: Serum proteomics
- Healthy Controls: Healthy volunteers
  Interventions: Other: Serum proteomics

INTERVENTIONS:
Other: Serum proteomics — magnetic bead-based fractionation coupled with matrix-assisted laser desorption/ionization-time-of-flight mass spectrometry
  Other Names: MB coupled with MALDI-TOF MS

SUMMARY:
No ideal serum biomarker currently exists for the early diagnosis of colorectal cancer (CRC). Therefore, it is urgent that accurate and reliable serum biomarkers be identified.

DETAILED DESCRIPTION:
Magnetic bead-based fractionation coupled with matrix-assisted laser desorption/ionization-time-of-flight mass spectrometry (MALDI-TOF MS) was used to screen serum samples from CRC patients and healthy controls.

ELIGIBILITY:
Patients with colorectal cancer

Inclusion criteria

* histologically confirmed colorectal cancer
* aged 18 years or older
* have provided written informed consent

Exclusion criteria

* refusal to participate

Healthy controls

Inclusion criteria

* no cancer history
* aged 18 years or older
* have provided written informed consent

Exclusion criteria

* refusal to participate
* have first-degree relative with a known history of colorectal cancer

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All of the CRC serum samples were obtained from patients with histologically confirmed colorectal cancer in the Department of General Surgery, Zhongshan Hospital, Fudan University, China. The control samples were collected from healthy volunteers.
Sampling Method: Probability Sample
Enrollment: 547 (Actual)
Dates: Start 2007-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Serum peptide mass fingerprinting (PMF) | 2010.03-2012.05 (2 years)
  Compare PMF of the colorectal caner group and control group, and then build the model to distinguish patients with colorectal cancer and controls

SECONDARY OUTCOMES:
Expressed peptide peaks | 2010.03-2012.05 (2 years)
  Find differentially expressed peptide peaks from the model and identify some ideal serum biomarkers for the early diagnosis of colorectal cancer

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Xu, M.D.,Ph.D., Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Villanueva J, Shaffer DR, Philip J, Chaparro CA, Erdjument-Bromage H, Olshen AB, Fleisher M, Lilja H, Brogi E, Boyd J, Sanchez-Carbayo M, Holland EC, Cordon-Cardo C, Scher HI, Tempst P. Differential exoprotease activities confer tumor-specific serum peptidome patterns. J Clin Invest. 2006 Jan;116(1):271-84. doi: 10.1172/JCI26022. PMID 16395409
- [Background] Wulfkuhle JD, Liotta LA, Petricoin EF. Proteomic applications for the early detection of cancer. Nat Rev Cancer. 2003 Apr;3(4):267-75. doi: 10.1038/nrc1043. PMID 12671665
- [Background] Cheng AJ, Chen LC, Chien KY, Chen YJ, Chang JT, Wang HM, Liao CT, Chen IH. Oral cancer plasma tumor marker identified with bead-based affinity-fractionated proteomic technology. Clin Chem. 2005 Dec;51(12):2236-44. doi: 10.1373/clinchem.2005.052324. Epub 2005 Oct 20. PMID 16239339
- [Background] Freed GL, Cazares LH, Fichandler CE, Fuller TW, Sawyer CA, Stack BC Jr, Schraff S, Semmes OJ, Wadsworth JT, Drake RR. Differential capture of serum proteins for expression profiling and biomarker discovery in pre- and posttreatment head and neck cancer samples. Laryngoscope. 2008 Jan;118(1):61-8. doi: 10.1097/MLG.0b013e31814cf389. PMID 18043497
- [Background] Rosenblatt KP, Bryant-Greenwood P, Killian JK, Mehta A, Geho D, Espina V, Petricoin EF 3rd, Liotta LA. Serum proteomics in cancer diagnosis and management. Annu Rev Med. 2004;55:97-112. doi: 10.1146/annurev.med.55.091902.105237. PMID 14746511